CLINICAL TRIAL: NCT03149874
Title: Accelerated Vaccination Schedule Against Hepatitis B Virus With Combined Hepatitis A and B Vaccine Among Hemodialysis Patients, Does it Works?
Brief Title: Accelerated Vaccination Schedule Against Hepatitis B Virus With Combined Hepatitis A and B Vaccine Among Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Collaborators: New Jeddah Clinic Hospital (Industry)
Responsible Party: Principal Investigator, Mahmoud Hamada imam, MD. - Lecturer at Internal Medicine Department- Faculty of Medicine, Benha University
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: BN-0517
Record Dates: First submitted 2017-05-08; First posted 2017-05-11 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Hepatitis B; Hemodialysis Complication
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Intervention Model Description: Patient seuentially randomized to either vaccine
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hepatitis B recombinant DNA vaccine (Active Comparator): Each Hepatitis B recombinant DNA vaccine vial contained 20 microgram of vaccine dose. Two vials will be intramuscularly injected one vial in each deltoid muscle on months zero, one, two and six.
  Interventions: Drug: Hepatitis B recombinant DNA vaccine
- Combined hepatitis A and B vaccine (Active Comparator): Each one-milliliter dose of vaccine contains 720 ELISA units of inactivated hepatitis A virus and 20 mcg of recombinant HBsAg protein. One dose of vaccine also contains 0.45 mg of aluminum. Two vials will be intramuscularly injected one vial in each deltoid muscle on on days zero, seven, and 21.
  Interventions: Drug: Combined hepatitis A and B vaccine

INTERVENTIONS:
Drug: Hepatitis B recombinant DNA vaccine — Hepatitis B recombinant DNA vaccine
  Arms: Hepatitis B recombinant DNA vaccine
Drug: Combined hepatitis A and B vaccine — Combined hepatitis A and B vaccine given to the patients
  Arms: Combined hepatitis A and B vaccine

SUMMARY:
The aim of this study is to examine the result of seroprotection using the accelerated vaccination schedule in vaccination of hemodialysis patient through using combined hepatitis A and B vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Age was above 18 years
* Hemodialysis patient
* All patients had undetectable hepatitis B virus surface antigen and antibody

Exclusion Criteria:

* A positive serum hepatitis B virus surface antigen and antibody
* patient received a previous course of hepatitis B virus vaccine

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2014-12-01 (Actual); Primary Completion 2017-04-30 (Actual); Study Completion 2017-05-01 (Actual)

PRIMARY OUTCOMES:
Hepatitis B virus Seroprotection after one month | one month after third dose of the vaccine
  Hepatitis B virus surface antibodies titer after one month
Hepatitis B virus Seroprotection after three months | three months after third dose of the vaccine
  Hepatitis B virus surface antibodies titer after three month

SECONDARY OUTCOMES:
Fever | 4 Days after each vaccination dose
  The proportion of fever among patients in both arms
Pain scale | 1 Hour after each vaccination dose
  Visual pain scale for pain from injection

IPD SHARING:
Plan to Share IPD: No